CLINICAL TRIAL: NCT03127904
Title: Pragmatic, Bayesian Adaptive Trial Comparing the Venfit System Against Standard Compressive Therapy in the Treatment of Venous Ulcers
Brief Title: Vein Fitness System vs Compressive Therapy for Venous Ulcers: a Bayesian Adaptive Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pró Circulação® (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Procirculacao1
Record Dates: First submitted 2017-03-24; First posted 2017-04-25 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Varicose Ulcer
Keywords: Varicose ulcer; Compressive therapy; Venous ulcer; Chronic venous disease
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Outcome evaluators and data scientists will be blinded regarding randomization. Blinding will be ensured by asking investigators at the end of the trial if investigators knew the arm to which each subject was going to be allocated prior to opening the envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vein Fitness (Experimental): Lymphomiokinetic exercises will be performed during a 1 hour period, with the patients in a supine position, legs elevated and properly positioned on a carpet; the knees will be mildly flexed to a comfortable point. The patients will put feet on the pedals of ankle extension/flexion device. The frequency will be around 15 to 20 cycles/minute, while the amplitude will be individually adjusted according to the range of movement of each patient. During the exercises, study personnel will manually drain the lower members.
  Compressive therapy will be applied as described in the control group arm.
  Care of the wound will be delivered as described in the control group arm.
  Interventions: Procedure: Vein Fitness; Procedure: Compressive therapy and wound care
- Control group (Active Comparator): Compressive therapy will be applied to both groups by properly trained personnel. Each layer of the compressive boot will have a 50% overlap, from the base to of the fingers to 3 cm bellow the popliteal fossa. The interface pressure used will be of at least 50mmHg in supine position.
  Wound care will be delivered to every individual in both groups, 1 or 2 times each week by a nurse certified in wound management, following the principles of maintenance of a moisturized surface between the wound and its cover. The nurse will also carry out mechanical wound debriding and biofilm removal.
  Interventions: Procedure: Compressive therapy and wound care

INTERVENTIONS:
Procedure: Vein Fitness — Vein fitness is a combination of whole-limb exercises, manual lymphatic drainage, and usual care (wound care and compressive therapy).
  Arms: Vein Fitness
Procedure: Compressive therapy and wound care — Compressive therapy consists in the application of pressure to the inferior limb. Investigators describe the specifics in the arm section.
  As previously described, a trained nurse will be in charge of keeping the wound healthy, verifying the surface is clean, debriding it, and removing biofilm from it.

SUMMARY:
The objective of this Bayesian Adaptive trial is to compare a control group versus a comprehensive ulcer healing protocol. The latter involves a combination of compressive therapy, miokinetic drainage and muscle strengthening for the entire lower extremity pump among patients with lower extremity venous ulcers. The investigators hypothesized that the combined therapy will have a higher closure rate as well as lower time to closure.

DETAILED DESCRIPTION:
This is a Bayesian adaptive, randomized, controlled, parallel, two-armed Bayesian adaptive trial. Patients diagnosed with varicose ulcers through Doppler ultrasonography will be recruited at the Pro Circulation Clinic of Angiology and Vascular Surgery, Brazil. The active group will be the Vein Fitness system, a multimodal intervention comprising exercise, lymphatic drainage, and compressive therapy, while the control group will be standard compressive therapy and regular wound care. The researchers will measure closure of the wounds and the closure rate as the primary outcomes. The study was designed in accordance with the CONSORT statement.

ELIGIBILITY:
Inclusion Criteria:

* Venous ulcers due to chronic venous disease assessed by color duplex scan (CDS) examination in standing position. Reflux will be assessed using CDS over a longitudinal vein through the manual compression of the calf in a distant position from the examined area. Reflux will be considered pathological if: >0.5 seconds (s) in the superficial venous system, or > 1.0 s in the deep system, or > 0.35 s in a perforator vein.

Exclusion Criteria:

* Investigators will exclude patients with ulcers from any other cause, including arterial insufficiency, with ankle-brachial pressure index (ABPI) < 0.8. Also will be excluded patients who use immunosuppressive and chemotherapy drugs, who have allergies to compression materials, and wheelchair users (due to the impossibility of performing the exercises).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-07-24 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Healing of venous ulcer. | 3 months
  Healing is defined as having the ulcer fully covered with scarring tissue.
Rate of ulcer closure | 3 months
  A ratio of the ulcer area and the time that it takes to close. Ulcer size will be measured using a standard protocol: First, we will photograph the wounds at a standard one meter distance having a ruler besides the lower extremity. The area of each wound will then be estimated through the Imagej software (National Institutes of Health) using a freehand drawing surrounding its border, with software calibration based on the pre-established dimensions of the background image. We will also assess a subset of 20 images by two independent observers to estimate inter-observer reliability.

SECONDARY OUTCOMES:
Time-to-closure | 3 months
  The time that it takes for an ulcer to close. Ulcer size will be measured using a standard protocol: First, we will photograph the wounds at a standard one meter distance having a ruler besides the lower extremity. The area of each wound will then be estimated through the Imagej software (National Institutes of Health) using a freehand drawing surrounding its border, with software calibration based on the pre-established dimensions of the background image. We will also assess a subset of 20 images by two independent observers to estimate inter-observer reliability.
Ankle range of motion | 3 months
  The angle that the ankle can reach as it moves. We will measure ankle range of motion through a goniometer. Specifically, passive ankle motion will be performed, with the fixed arm of the goniometer located on the leg axis, aligning the movable arm with the foot axis. We will perform all procedures in an office setting by trained physical therapists. A random group of patients will have the goniometry procedure performed twice by two independent physical therapists to assess the inter-observer reliability of these metrics.
Leg strength | 3 months
  The stand-up test will be used to measure the force of the inferior limb
Health-related quality of Life | 3 months
  Heath related quality of life will be assessed with a validated Portuguese version of the SF-36 (Short-Form Health Survey) tool.
Leg perimetry | 3 months
  Perimetry will be conducted at two different levels of the foot, and at five distinct levels of the leg, using a regular commercial tape. No pressure will be applied to these measurements to avoid affecting their precision. We will conduct the first-foot measurement five centimeters proximal to the base of the first proximal phalanx of the second toe, and the second measurement five centimeters proximal to the first measure. The first leg measurement will be performed five centimeters above the inferior border of the lateral malleolus, and then followed at every five centimeters to a total of six to eight measurements depending on the leg height.
Barthel Index | 3 months
  An ordinal scale used to measure performance in activities of daily living (ADL). Ten variables evaluating ADL and mobility are scored. Each item is rated in terms of whether the individual can perform the task independently, with some assistance, or is dependent on help based on observation (0=unable, 1=needs help, 2=independent). The final score is x 5 to get a number on a 100 point score. SScores of 0-20 indicate "total" dependency, 21-60 represents "severe" dependency, 61-90 indicate "moderate" dependency, and 91-99 indicates "slight" dependency.
Lawton-Brody Instrumental Activities of Daily Living (iADL) | 3 months
  Used to assess independent living skills of an individual and measures functional ability. Each item is rated trichotomously (1 = unable, 2 = needs assistance, 3 = independent) and the score is the sum of the responses. The higher the score, the greater the person's abilities.
Physical Activity Questionnaire (IPAQ) | 3 months
  IPAQ assesses physical activity undertaken across a comprehensive set of domains, including leisure-time physical activity, domestic and gardening (yard) activities, work-related physical activity, and transport-related physical activity. The score is obtained by the sum of the duration (in minutes) and frequency (days) for all the types of activities in all domains. A higher score represents a higher level of physical activity.
Interface Pressure (IP) | 3 months
  Defined as the pressure exerted by the compression system over the surface of skin.
Static Stiffness Index (SSI) | 3 months
  Defined as the difference between standing and resting pressure
Working Pressure Amplitude (WPA) | 3 months
  Considered as the difference between the lowest and highest interface pressure recorded during flexion and extension movements.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Matta, MD, Principal Investigator — Pró Circulação®
Locations (1):
- Pró-Circulação - Clinic of Angiology and Vascular Surgery, Xanxerê, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No